CLINICAL TRIAL: NCT01396798
Title: Validation of Vital Signs and Symptoms for the Diagnosis of Serious Infections in Children in a High Prevalent Setting: the Paediatric A&E.
Brief Title: Validation of Vital Signs and Symptoms for the Diagnosis of Serious Infections in Children in the Paediatric A&E.
Acronym: ERNIE3
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Jan Verbakel, Jan Verbakel, M.D., KU Leuven
Other Study IDs: S52996
Record Dates: First submitted 2011-07-18; First posted 2011-07-19 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Community-Acquired Infections; Respiratory Tract Infections; Sepsis; Urinary Tract Infections; Meningitis; Gastroenteritis
Keywords: serious infections; meningitis
MeSH Terms: conditions — Community-Acquired Infections; Respiratory Tract Infections; Sepsis; Urinary Tract Infections; Meningitis; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children with an acute illness: Children aged 1 month to 16 years of age, which attend the A&E department of UZLeuven with an acute illness episode of maximum 5 days.

SUMMARY:
Validation of Vital Signs and Symptoms for the Diagnosis of Serious Infections in Acutely Ill Children in a High Prevalent Setting: The Paediatric Accidents & Emergencies through prospective observational data collection concerning specific items from the clinical and technical examination in diagnosing serious infections, such as meningitis, sepsis, pneumonia, pyelonephritis, bronchiolitis with hypoxia. Eventually we will attempt to validate a vital signs and symptoms rule derived from multiple low to high prevalent settings of acutely ill children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 month to 16 years
* Acute illness episode of maximum 5 days

Exclusion Criteria:

* recent trauma
* neurological conditions
* intoxication
* psychiatric of behavioural disorders without a somatic cause
* acute exacerbation of a chronic condition (asthma, known immunodeficiency, diabetes, cystic fibrosis, etc)

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1 month to 16 years, attending the A&E department of the UZLeuven Hospital with an acute illness episode of maximum 5 days
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
serious infections: meningitis, sepsis, pneumonia, pyelonephritis, osteomyelitis and cellulitis, gastroenteritis with sever dehydration, complicated urinary tract infection and complicated viral airway infection with hypoxia. | within 24 hours after assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jan YJ Verbakel, M.D., Principal Investigator — KU Leuven
Locations (1):
- Dienst Algemene Kindergeneeskunde, Universitaire Ziekenhuizen Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Van den Bruel A, Haj-Hassan T, Thompson M, Buntinx F, Mant D; European Research Network on Recognising Serious Infection investigators. Diagnostic value of clinical features at presentation to identify serious infection in children in developed countries: a systematic review. Lancet. 2010 Mar 6;375(9717):834-45. doi: 10.1016/S0140-6736(09)62000-6. Epub 2010 Feb 2. PMID 20132979
- [Background] Van den Bruel A, Aertgeerts B, Bruyninckx R, Aerts M, Buntinx F. Signs and symptoms for diagnosis of serious infections in children: a prospective study in primary care. Br J Gen Pract. 2007 Jul;57(540):538-46. PMID 17727746